CLINICAL TRIAL: NCT00713128
Title: Prospective Evaluation of the Incidence of Nausea and Vomiting in Patients With Colorectal Cancer Receiving Irinotecan-based Therapy
Brief Title: Evaluation of the Incidence of Nausea and Vomiting in Patients With Colorectal Cancer Receiving Irinotecan-based Therapy
Status: Completed | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Paul J. Hesketh, M.D. Chief Division of Hematology/Oncology, Caritas St. Elizabeth's Medical Center of Boston
Other Study IDs: 00455
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer
Keywords: nausea vomiting colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study to determine how much nausea and or vomiting is caused by irinotecan-based chemotherapy in patients with colorectal cancer. Patients with colorectal cancer scheduled to receive their first cycle of an irinotecan-based chemotherapy regimen are eligible. Any chemotherapy agents administered in combination with irinotecan must have low-minimal potential to cause nausea and or vomiting. Examples of acceptable regimens would be irinotecan in combination with infusional fluorouracil and leucovorin (FOLFRI) with or without bevacizumab and irinotecan in combination with cetuximab. Patients who have received prior non-irinotecan-based chemotherapy are eligible providing they experienced no vomiting and no greater than mild nausea with their prior chemotherapy.

DETAILED DESCRIPTION:
Irinotecan is a camptothecin analog which exerts its cytotoxic effects by forming a covalent complex with topoisomerase I and DNA, resulting in inhibition of DNA re-ligation, accumulation of DNA double strand breaks and apoptotic cell death (1). Irinotecan is FDA approved for use in the front-line and second-line treatment of colorectal cancer. It has also demonstrated activity in a variety of other non-hematologic tumors. The recently updated ASCO antiemetic guidelines characterize irinotecan as having moderate emetic risk. (2). However, the emetogenic potential of this agent has been poorly characterized and there are no published prospective trials with emesis as a primary-end point. In addition there is a complete paucity of information on the potential of irinotecan to induce emesis beyond the first day after chemotherapy, so-called delayed emesis. Best characterized following cisplatin, delayed emesis is also associated with a number of other chemotherapy agents that similar to irinotecan appear to be moderately emetogenic such as carboplatin, cyclophosphamide and doxorubicin. Antiemetic prophylaxis for delayed emesis following irinotecan is not routinely prescribed at the present time. Prospectively obtained information on the potential of irinotecan to cause delayed emesis would be helpful in guiding appropriate antiemetic practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer receiving irinotecan in combination with infusional fluorouracil and leucovorin (FOLFRI) with or without bevacizumab or irinotecan in combination with cetuximab
* All patients will receive the following standard antiemetic regimen prior to chemotherapy:
* Dexamethasone 8 mg PO/IV
* An approved dose of a 5HT3 receptor antagonist. Ondansetron 8mg IV or 24mg PO Dolasetron 100mg IV/PO Granisetron 1 mg IV or 2mg PO Use of palonosetron will be excluded on this trial No routine prophylaxis for delayed emesis will be given. Patients will be instructed in the use of rescue antiemetics if needed.
* Minimum age of 18 years.
* Premenopausal patients must demonstrate a negative serum or urine pregnancy test prior to receiving chemotherapy.
* ECOG performance status of 0-2 (Appendix A)
* Execution of written informed consent

Exclusion Criteria:

* Patients with history of moderate-severe nausea or any vomiting with prior chemotherapy including irinotecan based chemotherapy.
* Concomitant use of any drug with potential antiemetic efficacy (Appendix B) 24 hours before chemotherapy and during the 120 hour study period. Chronic use (more than 2 weeks) of benzodiazepines is allowed.
* Vomiting, retching or nausea (NCI > 1) in the 24 hours preceding chemotherapy
* Palliative surgery < 2 weeks from study entry
* Concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer receiving Irinotecan based therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
frequency of delayed emesis (vomiting/retching) | days 2 - 5

SECONDARY OUTCOMES:
Freq. of mild-severe nausea D 2-6 Freq. use of antiemetics D 2-6, Pts.with complete response(no emesis/use of rescue antiemtics)D 1, Pts. with total control (no:emesis,nausea, use of rescue antiemetics)D 2-6, Overall satisfaction | 120 hours (days 1 thru 5)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Hesketh, M.D., Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- Caritas St. Elizabeth Medical Center, Brighton, Massachusetts, United States